CLINICAL TRIAL: NCT02836210
Title: 27-gauge Vitrectomy Wound Integrity: a Prospective, Randomized Trial Comparing Angled Versus Straight Entry in Fluid-filled Vitrectomized Eyes
Brief Title: 27-gauge Vitrectomy Wound Integrity: a Prospective, Randomized Trial Comparing Angled Versus Straight Entry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Dr. Carl D. Regillo, MD, Wills Eye
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: WEH IRB# 15-514
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Epiretinal Membrane
Keywords: 27-gauge Pars plana vitrectomy
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angled incision (Active Comparator): Patients in this arm will undergo 27-gauge vitrectomy wound construction using angled (tunnel-like) incisions for trocar entry.
  Interventions: Device: 27-gauge vitrectomy wound construction
- Straight Incision (Active Comparator): Patients in this arm undergo 27-gauge vitrectomy wound construction using straight (perpendicular) incisions for trocar entry.
  Interventions: Device: 27-gauge vitrectomy wound construction

INTERVENTIONS:
Device: 27-gauge vitrectomy wound construction — Conventional, 3-port pars plana vitrectomy with membrane peeling is performed for epiretinal membrane indication. Angled and straight trocar entry will be directly compared.

SUMMARY:
To prospectively compare clinical outcomes using straight (perpendicular) versus angled trocar insertion during 27 gauge pars plana vitrectomy surgery for epiretinal membrane

Primary Endpoints:

Sclerotomy suture rates and incidence of suture blebs at the end of 27 gauge MIVS.

Secondary Endpoints:

Rate of postoperative wound-related complications such as hypotony, choroidal detachments, endophthalmitis, and sclerotomy-related retinal tears with a minimum follow-up of 30 days.

DETAILED DESCRIPTION:
Microincision vitrectomy surgery (MIVS) has largely replaced use of conventional, 20-gauge vitrectomy, offering more rapid visual recovery, decreased postoperative pain and inflammation, and reduced surgical time with use of smaller diameter instruments1. Most recently, 27 gauge vitrectomy instrumentation has been introduced2, offering an additional small gauge option to the currently available 23, 25, or 25+ gauge systems.

Initial experience with small gauge MIVS yielded mixed results, with early reports noting increased rates of wound-related postoperative complications including hypotony, choroidal detachments, endophthalmitis, and sclerotomy-related retinal tears3,4. However, with more experience and instrument modifications, outcomes with MIVS improved1,3. In a 2010 Ophthalmic Technology Assessment report by the American Academy of Ophthalmology, outcomes of MIVS were found comparable to that of 20 gauge vitrectomy benchmarks5.

Prior studies have established that a two-stage, angled incision results in improved wound integrity with 23, 25, and 25+ MIVS systems6,7, helping to prevent complications such as post-operative endophthalmitis and hypotony. However, in the two clinical series describing outcomes of 27 gauge MIVS, a one-stage, perpendicular wound construction was performed without complication in a series of 31 patients2,8. Thus far, direct comparison between wound construction techniques (one-stage, perpendicular or two-stage, angled) has not been evaluated.

The purpose of this study is to prospectively compare clinical outcomes using straight, one-stage (perpendicular) versus angled, two-stage trocar insertion during 27 gauge minimally invasive vitrectomy surgery (MIVS). The design of the study will be a randomized, clinical trial. Primary outcomes will be sclerotomy suture rates and incidence of suture blebs at the end of 27 gauge MIVS surgery for epiretinal membrane and macular pucker indications (no air or gas tamponade). Secondary endpoints will include rate of postoperative wound-related complications such as hypotony, choroidal detachments, endophthalmitis, and sclerotomy-related retinal tears with a minimum of 30 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old undergoing 27 gauge vitrectomy surgery with membrane peel for epiretinal membrane
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* History of previous vitrectomy surgery in the study eye.
* History of previous ocular surgery other than cataract extraction in the study eye.
* Requirement of an air or gas (SF6, C3F8) bubble at the conclusion of 27 gauge MIVS surgery.
* Aphakia, ACIOL, unstable PCIOL, and/or lenticular or zonular instability.
* Glaucoma requiring IOP lowering medications.
* Pre-existing ocular inflammation/uveitis.
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either require medical or surgical intervention during the 12 week study period to prevent or treat visual loss that might result from that condition. Examples include infectious conjunctivitis, keratitis, and/or scleritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Rate of sclerotomy site suturing and suture bleb formation | Minimum follow-up 30 days.

SECONDARY OUTCOMES:
Rate of post-operative, wound related complications | Minimum follow-up of 30 days
  Rate of complications including hypotony, choroidal detachment, and endophthalmitis
Change in mean intraocular pressure | Minimum follow-up of 30 days
  Measured in mm Hg by tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Carl D Regillo, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thompson JT. Advantages and limitations of small gauge vitrectomy. Surv Ophthalmol. 2011 Mar-Apr;56(2):162-72. doi: 10.1016/j.survophthal.2010.08.003. Epub 2011 Jan 14. PMID 21236459
- [Background] Oshima Y, Wakabayashi T, Sato T, Ohji M, Tano Y. A 27-gauge instrument system for transconjunctival sutureless microincision vitrectomy surgery. Ophthalmology. 2010 Jan;117(1):93-102.e2. doi: 10.1016/j.ophtha.2009.06.043. Epub 2009 Oct 31. PMID 19880185
- [Background] Spirn MJ. Comparison of 25, 23 and 20-gauge vitrectomy. Curr Opin Ophthalmol. 2009 May;20(3):195-9. doi: 10.1097/ICU.0b013e328329eaea. PMID 19390437
- [Background] Chen E. 25-Gauge transconjunctival sutureless vitrectomy. Curr Opin Ophthalmol. 2007 May;18(3):188-93. doi: 10.1097/ICU.0b013e328133889a. PMID 17435424
- [Background] Recchia FM, Scott IU, Brown GC, Brown MM, Ho AC, Ip MS. Small-gauge pars plana vitrectomy: a report by the American Academy of Ophthalmology. Ophthalmology. 2010 Sep;117(9):1851-7. doi: 10.1016/j.ophtha.2010.06.014. PMID 20816248
- [Background] Rizzo S, Barca F, Caporossi T, Mariotti C. Twenty-seven-gauge vitrectomy for various vitreoretinal diseases. Retina. 2015 Jun;35(6):1273-8. doi: 10.1097/IAE.0000000000000545. No abstract available. PMID 25946694
- [Background] Gupta OP, Maguire JI, Eagle RC Jr, Garg SJ, Gonye GE. The competency of pars plana vitrectomy incisions: a comparative histologic and spectrophotometric analysis. Am J Ophthalmol. 2009 Feb;147(2):243-250.e1. doi: 10.1016/j.ajo.2008.08.025. Epub 2008 Oct 23. PMID 18947818
- [Background] Teixeira A, Rezende FA, Salaroli C, Souza N, Sousa BA, Allemann N. In vivo comparison of 23- and 25-gauge sutureless vitrectomy incision architecture using spectral domain optical coherence tomography. J Ophthalmol. 2013;2013:347801. doi: 10.1155/2013/347801. Epub 2013 Mar 4. PMID 23533705